CLINICAL TRIAL: NCT04607109
Title: Neurodevelopmental Assessment and Parents Feelings at 7-8 Years of Age for Prematurely Born Children Involved in the Réseau Périnatal Lorrain Follow-up Program
Brief Title: Long-term Neurodevelopmental Disorders of Prematurely Born Children and Parental Experience
Acronym: PREMA7
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI166
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Neurodevelopmental Abnormality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thanks to the evolution in knowledge and technical advances in premature newborn intensive care, the survival of very premature infants is now possible. However, prognosis remain sometimes uncertain.

In 2011, the Epipage 2 study showed a significant improvement as compared with the 1997 Epipage1 study with a decrease in mortality and an increase of the survival rate without severe morbidity of 14% for preterm babies born between 25 and 29 weeks and 6% for babies born between 30 and 31 weeks.

However, surviving babies without initial major deficiencies, may later show problems in terms of growth, sensory - motor and/or neuro-psychologic development. This untoward evolution lead to social and family interaction disorders and school difficulties.

In this context, a perinatal care network was created for each Region in France, making it possible to take care of these vulnerable children early on and all along their development. A retrospective study will evaluate 97 pre-term babies born before 33 weeks in 2012 and who are taken care of at Nancy as part of the Lorraine regional network program "Rafael" until they are 7 years old.

The objective is to evaluate objectively the neurocognitive and school abilities of these children at the age of 7.

At 8 years of age, a secondary measure of outcome will be the impact of the eventual neurocognitive consequences on the quality of their family life, on the behavior of the child and the parents' feelings. This way more options to improve the way they are taken care of will be available.

ELIGIBILITY:
Inclusion Criteria:

* all children prematurely born between 24 and 33 completed week during 2012
* and involved in the Lorraine Perinatal Follow-up program at 7 years old

Exclusion Criteria:

* Children not able to respond to the EDA evaluation

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born prematurely (< 33SA) in 2012 and followed up in the RAFAEL network 7 years of age
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
EDA score (Evaluation Des fonctions cognitives et des Apprentissages) | 7 years old
  Evaluation of learning ability by a standardized score (ranging from 15 in maths to 65 in reading, the higher score being the better)

SECONDARY OUTCOMES:
RAFAEL follow-up questionnaire reply of parents | 8 years old
  Questionnaire on parents feelings (with 4 levels from no impact to heavy disturbances of the family life)

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Hospital CHRU, Nancy, France